CLINICAL TRIAL: NCT05645354
Title: SmokefreeSGM, A Text-based Smoking Cessation Feasibility Trial for Sexual and Gender Minority Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Irene Tami-Maury, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-22-0717; K22CA237639 (NIH)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: lesbian, gay, bisexual, transgender, queer (LGBTQ)
MeSH Terms: conditions — Smoking Cessation; Homosexuality, Female; Homosexuality; Bisexuality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmokefreeSGM (Experimental)
  Interventions: Behavioral: SmokefreeSGM
- SmokefreeTXT (Active Comparator)
  Interventions: Behavioral: SmokefreeTXT

INTERVENTIONS:
Behavioral: SmokefreeSGM — Participants will be enrolled in a text-based smoking cessation program specifically designed to respond to the needs of LGBTQ+ smokers.
  Arms: SmokefreeSGM
Behavioral: SmokefreeTXT — Participants will be enrolled in a text-based smoking cessation program specifically designed to respond to the needs of the general population
  Arms: SmokefreeTXT

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of Smokefree Sexual and Gender Minority (SGM), an SGM-tailored version of the SmokefreeTXT text messaging program

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as an LGBTQ+ individual
* Currently live in the United States
* Have smoked at least 100 cigarettes in their lifetime, smoke every day, and smoke greater than or equal to 5 cigarettes a day
* Are willing to quit smoking in the next 15 days
* Have a cell phone number with an unlimited short message service (SMS) plan
* Have a positive cotinine saliva test to indicate their smoking status

Exclusion Criteria:

* Have a prepaid cell phone plan (pay-as-you-go plan)
* Have a cell phone number that does not work and/or is registered to someone else
* Have inadequate equipment/devices (i.e., webcam, speakers, mic) for participating in telehealth sessions via Microsoft Teams, Webex, or Zoom AND cannot meet in-person
* Pregnant or breastfeeding persons (nicotine patches are not generally recommended to this groups since nicotine can affect fetal and neonatal brain development)
* Contraindication for nicotine patches. Absolute contraindications include: severe eczema or serious skin conditions, allergy to nicotine patches, pregnancy, breastfeeding, heart attack in the past 2 months, ongoing angina, peptic ulcer disease, arrhythmia, or uncontrolled blood pressure. Potential contraindications include: stroke in the past 6 months, insulin therapy, and a current diagnosis of liver, kidney, or heart disease. Study participants reporting a potential contraindication will require approval from their primary care provider and/or other treating physician (e.g., psychiatrist) to use nicotine patches. If the request is denied or not returned in 2 weeks, potential study participants will be excluded from the study.
* Current use of tobacco cessation medications
* Enrollment in another smoking cessation study
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as a lesbian, gay, bisexual, transgender or queer individual
Enrollment: 100 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tami-Maury, DMD, DrPH, MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tundealao S, Oubda MC, Klaff R, Reininger B, McNeill L, Tami-Maury I. Pragmatic recruitment strategies for a text-based smoking cessation intervention for sexual and gender minority groups. Discov Public Health. 2025;22(1):743. doi: 10.1186/s12982-025-01117-0. Epub 2025 Nov 24. PMID 41306822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 217 participants screened, 100 participants met all inclusion criteria, were enrolled and randomized.
Period: Overall Study
Arm/Group | SmokefreeSGM | SmokefreeTXT
Started | 50 | 50
Completed 1 Month Follow up | 35 | 34
Completed 3 Month Follow up | 22 | 20
Completed 6 Month Follow up | 19 | 16
Completed | 19 | 16
Not Completed | 31 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SmokefreeTXT | SmokefreeSGM | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.7) | 38.2 (12.2) | 41.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 20 | 23 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 29 | 31 | 60
  Non-Hispanic Black | 10 | 15 | 25
  Hispanic | 6 | 4 | 10
  Other | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Sexual Orientation [Count of Participants; unit: Participants]
  Gay Male/Bisexual Male | 20 | 17 | 37
  Lesbian/Gay Woman/ Bisexual Female | 24 | 26 | 50
  Others (pansexual, queer, unsure) | 6 | 7 | 13
Work Status [Count of Participants; unit: Participants]
  Working | 29 | 28 | 57
  Not Working | 21 | 22 | 43
Level of Education [Count of Participants; unit: Participants]
  less than or equal to High school | 9 | 13 | 22
  Technical/vocational degree/ Completed some college | 28 | 19 | 47
  Bachelor's/ master's /associate degree | 13 | 18 | 31
Marital Status [Count of Participants; unit: Participants]
  Single/Separate/Divorced/Widowed | 36 | 36 | 72
  Married/Living with significant other | 14 | 14 | 28
Children in household [Count of Participants; unit: Participants]
  No | 38 | 38 | 76
  Yes | 12 | 12 | 24
Number of Participants who live with other smokers [Count of Participants; unit: Participants] | 19 | 16 | 35
Number of times participants tried to quit smoking [Count of Participants; unit: Participants]
  Never tried | 2 | 4 | 6
  Between 1 and 10 times | 35 | 38 | 73
  More than 10 times | 13 | 8 | 21
Age at smoking initation [Mean (Standard Deviation); unit: years] | 15.3 (2.7) | 14.3 (3.3) | 14.8 (3.1)
Nicotine dependence as assessed by the Fagerstrom Test for Nicotine Dependence [Count of Participants; unit: Participants] — The Fagerström Test for Nicotine Dependence (FTND) is a standard instrument for assessing the intensity of physical addiction to nicotine. The total score ranges from 0 to 10. Participants were categorized as mild (between 0 and 3), moderate(between 4 and 6) or severe (greater than 7) nicotine dependence based on their FTND score.
  Participants
    mild dependance on nicotine | 11 | 11 | 22
    moderate dependance on nicotine | 33 | 22 | 55
    severe dependance on nicotine | 6 | 17 | 23
E-cigarette Dependence as assessed by Penn State E-cigarette Dependence Index [Count of Participants; unit: Participants] — The Penn State E-cigarette Dependence Index is a standard instrument for assessing e-cigarette dependence. The total score ranges from 0 to 20. Participants were categorized as Not dependent (between 0 and 3), Low dependence (between 4 and 8), medium dependence (between 9 and 12, or high dependence (greater than 13) based off their score. Population: Data for this outcome measure was collected for only the participants who smoke electronic cigarettes.
  Participants
    number analyzed (Participants) | 27 | 13 | 40
    Not Dependent | 8 | 4 | 12
    Low dependence | 6 | 3 | 9
    medium dependence | 5 | 2 | 7
    high dependence | 8 | 4 | 12
Number of participants who smoke electronic cigarettes [Count of Participants; unit: Participants] | 27 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Number of Participants Recruited for the Study
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Screened: All Participants Screened
Arm/Group | All Participants Screened
Number analyzed (Participants) | 217
Participants | 100

2. Primary Outcome: Feasibility as Assessed by Number of Participants That Completed Month 1 Visit
Time Frame: end of month 1
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeSGM | SmokefreeTXT
Number analyzed (Participants) | 50 | 50
Participants | 35 | 34

3. Primary Outcome: Feasibility as Assessed by Number of Participants That Completed Month 3 Visit
Time Frame: end of month 3
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeSGM | SmokefreeTXT
Number analyzed (Participants) | 50 | 50
Participants | 22 | 20

4. Primary Outcome: Feasibility as Assessed by Number of Participants That Completed Month 6 Visit
Time Frame: end of month 6
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeSGM | SmokefreeTXT
Number analyzed (Participants) | 50 | 50
Participants | 19 | 16

5. Primary Outcome: Acceptability as Assessed by Number of Participants Who Completed Qualitative Interviews
Time Frame: 6 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeSGM | SmokefreeTXT
Number analyzed (Participants) | 19 | 16
Participants | 16 | 9

6. Secondary Outcome: Number of Participants That Quit Smoking
Time Frame: 1 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeTXT | SmokefreeSGM
Number analyzed (Participants) | 34 | 35
Participants | 18 | 15

7. Secondary Outcome: Number of Participants That Quit Smoking
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeTXT | SmokefreeSGM
Number analyzed (Participants) | 20 | 22
Participants | 7 | 8

8. Secondary Outcome: Number of Participants That Quit Smoking
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | SmokefreeTXT | SmokefreeSGM
Number analyzed (Participants) | 16 | 19
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | SmokefreeSGM | SmokefreeTXT
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SmokefreeSGM (N=50) | SmokefreeTXT (N=50)
Nausea (General disorders) | 0 | 1
Palpitations (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05645354/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05645354/ICF_001.pdf